CLINICAL TRIAL: NCT03289780
Title: An Observational Study Assessing the Clinical Effectiveness of VeriStrat and Validating Immunotherapy Tests in Subjects With Non-Small Cell Lung Cancer
Brief Title: Clinical Effectiveness Assessment of VeriStrat® Testing and Validation of Immunotherapy Tests in NSCLC Subjects
Acronym: INSIGHT
Status: Active, not recruiting | Type: Observational
Sponsor: Biodesix, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BDX-00146
Record Dates: First submitted 2017-08-16; First posted 2017-09-21 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to collect information about how a doctor uses the results of the VeriStrat® blood test to guide treatment for non-small cell lung cancer (NSCLC) patients. Understanding how VeriStrat test results influence doctors' decisions and patients' outcomes may help doctors to better treat NSCLC in the future. This study will also look to establish whether new investigational tests can help better predict the effectiveness of certain medications for certain patients. These new investigational tests are only for research purposes at this time.

DETAILED DESCRIPTION:
The primary purpose of this observational study is to assess the physician's clinical practice patterns while using VeriStrat testing in subjects with NSCLC whose tumors are epidermal growth factor receptor (EGFR) wild-type (negative) or have unknown EGFR mutational status. This study will also attempt to further validate that VeriStrat test results stratify subjects by clinical outcomes in the real world, uncontrolled clinical setting while exploring whether certain therapeutic approaches may yield opportunities for further study.

Predictive tests that aid physician therapeutic decision making are critical for optimizing subject outcomes while minimizing toxicity and associated treatment costs. This study will provide data for the validation of immunotherapy tests currently being developed. Immunotherapy mechanisms are dependent upon the interactions between the tumor, tumor microenvironment, and the patient immune system. As such, a successful predictive test will reflect the complex interplay between tumor and host. The multivariate tests from Biodesix have the advantage of being able to assess this complex biology.

The information gained from this research will not only guide the adoption of the VeriStrat test and inform medical decision making, including treatment choice, but will allow the validation of additional mass-spectrometry-based proteomic tests.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 years of age or older at time of signing informed consent form (ICF).
2. A diagnosis of NSCLC.
3. Subject is willing to provide serum samples for VeriStrat testing.
4. EGFR mutation status wild-type (negative) or a tested unknown.
5. For subjects with untested/unknown EGFR status only: The subject must be willing to provide blood samples for GeneStrat testing.
6. Subject is willing to provide serum samples for research, understanding that no test results will be made available either to the subject or the treating physician.
7. Subject is able to read and understand the ICF and agrees to comply with study procedures and requirements.

Exclusion Criteria:

1. Subject's ability to understand the requirements of the protocol or to provide informed consent is impaired or subject is unwilling to comply with the protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any Subject with Non-Small Cell Lung Cancer (NSCLC) at all stages with any histology.
Sampling Method: Non-Probability Sample
Enrollment: 5006 (Actual)
Dates: Start 2016-04-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Physician Treatment Patterns Description | 3 years
  Physician Treatment patterns Description: To describe physician treatment patterns pre and post-veriStrat testing. Describe the impact of the VeriStrat test results on treatment decisions, including but not limited to: percentage change in treatment decision, differences in chosen treatments between patients classified as VeriStrat good and those classified as VeriStrat Poor. Change in percentage of patients receiving systemic therapy or supportive therapies only.

SECONDARY OUTCOMES:
Immunotherapy Stratification by Overall Survival | 3 years
  To determine whether immunotherapy test(s) stratify immunotherapy-treated subjects by overall survival.
Immunotherapy Stratification by Progression-Free Survival | 3 years
  To determine whether immunotherapy test(s) stratify immunotherapy-treated subjects by progression-free survival.
VeriStrat Poor vs. Good Outcomes | 3 years
  To compare progression free survival (PFS) and overall survival (OS) outcomes between those classified as VeriStrat-Poor and VeriStrat-Good.
Platinum-based therapy outcomes in VeriStrat Poor vs. Good subjects. | 3 years
  To compare outcomes in subjects classified as VeriStrat-Poor and VeriStrat-Good and treated with platinum-based therapy.
Immunotherapy outcomes in VeriStrat Poor vs. Good subjects. | 3 years
  To compare outcomes in subjects classified as VeriStrat-Poor and VeriStrat-Good and treated with immunotherapy.
Single agent chemotherapy outcomes in VeriStrat Poor vs. Good Subjects | 3 years
  To compare outcomes in subjects classified as VeriStrat-Poor and VeriStrat-Good and treated with single agent chemotherapy.
VeriStrat label changes over time. | 3 years
  To compare the longitudinal changes in VeriStrat classification over the course of the study

OTHER OUTCOMES:
Determination of Immunotherapy tests ability to stratify subjects based on treatment. | 3 years
  To determine whether immunotherapy test(s) stratify subjects treated with chemotherapy or targeted therapies by outcome.
Correlation between the VeriStrat test and Immunotherapy tests. | 3 years
  To observe the correlation between VeriStrat classification and immunotherapy test(s) classification at baseline and longitudinally.
Longitudinal changes in Immunotherapy tests. | 3 years
  To describe the longitudinal changes in immunotherapy test classification over the course of the study.
Stratification of Immunotherapy Test(s) | 3 years
  To determine whether immunotherapy test(s) stratify immunotherapy-treated subjects by other clinically meaningful factors or endpoints.
Changes in GeneStrat | 3 years
  To observe changes in GeneStrat status across lines of therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Steve Springmeyer, MD, Principal Investigator — Biodesix, Inc.
Locations (42):
- United States (42):
  - Oncology Specialties, PC; Clearview Cancer Institute, Huntsville, Alabama
  - Lewis & Faye Manderson Cancer Center at DCH Regional Medical Center, Tuscaloosa, Alabama
  - Highlands Oncology Group, Fayetteville, Arkansas
  - St. Bernards Cancer Center Hematology / Oncology, Jonesboro, Arkansas
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Boca Raton Regional Hospital -Lynn Cancer Institute, Boca Raton, Florida
  - Lake City Cancer Care, LLC, Lake City, Florida
  - South Eastern Regional Medical Center, Newnan, Georgia
  - Summit Cancer Care, Savannah, Georgia
  - South Georgia Medical Center, Valdosta, Georgia
  - Edward-Elmhurst Healthcare, Naperville, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Franciscan Health Woodland Cancer Center, Michigan City, Indiana
  - Ponchartrain Cancer Center, Covington, Louisiana
  - Christus Health, Shreveport, Louisiana
  - North Mississippi Medical Center - Hematology and Oncology Clinic, Tupelo, Mississippi
  - Central Care Cancer Center, Bolivar, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - Mercy Medical, Springfield, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Essex Oncology, Belleville, New Jersey
  - New York Oncology Group, Albany, New York
  - Clinical Research Associates, Lake Success, New York
  - NYU Laura & Isaac Perlmutter Cancer Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Southeastern Medical Oncology, Goldsboro, North Carolina
  - Leo W. Jenkins Cancer Center - East Carolina University, Greenville, North Carolina
  - Hematology and Oncology Associates - Mercy Medical Center, Canton, Ohio
  - Tri-County Hematology & Oncology Associates, Massillon, Ohio
  - Oregon Oncology Specialists (QCCA), Salem, Oregon
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Bon Secours St. Francis Cancer Center, Greenville, South Carolina
  - Arlington Cancer Center, Arlington, Texas
  - JPS Health Network, JPS Center for Cancer Care, Fort Worth, Texas
  - The Center for Cancer and Blood Disorders, Fort Worth, Texas
  - Scott & White Memorial Hospital and Clinic, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Virginia Cancer Institute, Richmond, Virginia
  - Peace Health, Bellingham, Washington
  - Northwest Medical Specialties, PLLC, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akerley WL, Arnaud AM, Reddy B, Page RD. Impact of a multivariate serum-based proteomic test on physician treatment recommendations for advanced non-small-cell lung cancer. Curr Med Res Opin. 2017 Jun;33(6):1091-1097. doi: 10.1080/03007995.2017.1301903. Epub 2017 Mar 16. PMID 28277859
- [Background] Grossi F, Rijavec E, Genova C, Barletta G, Biello F, Maggioni C, Burrafato G, Sini C, Dal Bello MG, Meyer K, Roder J, Roder H, Grigorieva J. Serum proteomic test in advanced non-squamous non-small cell lung cancer treated in first line with standard chemotherapy. Br J Cancer. 2017 Jan 3;116(1):36-43. doi: 10.1038/bjc.2016.387. Epub 2016 Nov 29. PMID 27898657
- [Derived] Rich P, Mitchell RB, Schaefer E, Walker PR, Dubay JW, Boyd J, Oubre D, Page R, Khalil M, Sinha S, Boniol S, Halawani H, Santos ES, Brenner W, Orsini JM, Pauli E, Goldberg J, Veatch A, Haut M, Ghabach B, Bidyasar S, Quejada M, Khan W, Huang K, Traylor L, Akerley W. Real-world performance of blood-based proteomic profiling in first-line immunotherapy treatment in advanced stage non-small cell lung cancer. J Immunother Cancer. 2021 Oct;9(10):e002989. doi: 10.1136/jitc-2021-002989. PMID 34706885
- See also: Sponsor Website — http://www.biodesix.com

DOCUMENTS (2):
  • Study Protocol (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT03289780/Prot_003.pdf
  • Informed Consent Form (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT03289780/ICF_002.pdf